CLINICAL TRIAL: NCT03455439
Title: Risk Factors of Outcomes Associated With Disease Progression in Patients With Atrial Fibrillation and Heart Failure (HF) Who Are Receiving a Direct Oral Anticoagulant (Rivaroxaban)
Acronym: FARAONIC
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 19584
Record Dates: First submitted 2018-02-04; First posted 2018-03-06 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rivaroxaban: Adult patients diagnosed with Atrial Fibrilation and Heart Failure who started treatment with rivaroxaban at least 4 months prior to inclusion
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — As prescribed by the treating physician

SUMMARY:
Evaluation of the risk factors associated with Heart Failure (HF) worsening (measured by hospitalizations and emergency visits because of HF exacerbations) in Spanish patients with Atrial Fibrilation and HF treated with rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged 18 years or older.
* Patients with a diagnosis of nonvalvular Atrial Fibrilation (AF).
* Patients with a diagnosis of chronic Heart Failure, New York Heart Association (NYHA) class I-IV HF with preserved Ejection Fraction (HFpEF), HF with reduced EF (HFrEF) or HF with mid-range EF (HFmrEF).
* Patients receiving antithrombotic treatment because of AF, with rivaroxaban since at least 4 months before entering the study.
* Patients who have been given appropriate information about the study objectives and procedures and with the mental and physical capacity to give their informed consent to participate in the study.

Exclusion Criteria:

* Patients participating in a research program which involves some intervention beyond clinical practice.
* Patients who started rivaroxaban after the start of the inclusion period.
* Patients with significate mitral stenosis or other heart valvular diseases that requires or have needed specific treatment (prosthesis or valvuloplasty).
* Patients with severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Atrial Fibrilation and Heart Failure who started treatment with rivaroxaban at least 4 months prior to inclusion that attend the Cardiology Units or Internal Medicine Units at Spanish hospitals and private clinics.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Time from the baseline visit to the first hospitalization or admission to emergency services due to a Heart Failure exacerbation | Up to 24 months or early termination

SECONDARY OUTCOMES:
Date of death | Up to 24 months or early termination
Date of all hospitalizations or admissions to emergency service | Up to 24 months or early termination
  due to a HF exacerbation or all cause

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Background] Gomez Doblas JJ, Cepeda-Rodrigo JM, Agra Bermejo R, Blanco Labrador E, Blasco MT, Carrera Izquierdo M, Lekuona I, Recio Mayoral A, Rafols C, Manito N. Outcomes and factors associated with mortality in patients with atrial fibrillation and heart failure: FARAONIC study. Clin Cardiol. 2023 Nov;46(11):1390-1397. doi: 10.1002/clc.24106. Epub 2023 Aug 18. PMID 37596723
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/